CLINICAL TRIAL: NCT00910429
Title: Long-term Extension, Multicentre, Multi-international Study to Evaluate the Safety and Tolerability of Oral BAY63-2521 (1mg, 1.5 mg, 2.0 mg, 2.5 mg Tid) in Patients With Chronic Thromboembolic Pulmonary Hypertension (CTEPH).
Brief Title: BAY63-2521 - Long-term Extension Study in Patients With Chronic Thromboembolic Pulmonary Hypertension
Acronym: CHEST-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11349; 2008-003539-19 (EudraCT Number)
Record Dates: First submitted 2009-05-27; First posted 2009-05-29 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Hypertension
Keywords: Chronic thromboembolic Hypertension; PH; soluble Guanylate Cyclase Stimulator; sGC
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — BAY63-2521 - 1 mg tid - 2,5 mg tid orally until end of study

SUMMARY:
Patients who have completed the 16 weeks treatment of the CHEST-1 trial (study number 11348) will be asked to participate in this long term extension study with BAY63-2521. The aim of the long term study is to collect additional information to evaluate the safety and tolerability of BAY63-2521. Patients will be treated with open label medication on their individual optimal dose between 0,5 mg - 2,5 mg tid.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed 16 weeks of treatment in the double blind trial CHEST 1

Exclusion Criteria:

* Patients who have an ongoing serious adverse event from CHEST 1 that is assessed as related to BAY63-2521 are not allowed to participate in the extension trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (71):
- United States (8):
  - La Jolla, California
  - Sacramento, California
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dallas, Texas
- Corrientes, Argentina
- Prahran, Victoria, Australia
- Vienna, Austria
- Belgium (2):
  - Bruxelles - Brussel
  - Leuven
- Brazil (3):
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
  - Rio de Janeiro
- Canada (5):
  - Calgary, Alberta
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- China (2):
  - Beijing
  - Shanghai
- Prague, Czechia
- Aarhus N, Denmark
- France (4):
  - Brest
  - Le Kremlin-Bicêtre
  - Rouen
  - Vandœuvre-lès-Nancy
- Germany (10):
  - Heidelberg, Baden-Wurttemberg
  - München, Bavaria
  - Würzburg, Bavaria
  - Giessen, Hesse
  - Hanover, Lower Saxony
  - Cologne, North Rhine-Westphalia
  - Homburg, Saarland
  - Dresden, Saxony
  - Leipzig, Saxony
  - Hamburg
- Rabin Medical Center - Beilinson Campus, Petah Tikva, Israel
- Pavia, Lombardy, Italy
- Japan (11):
  - Nagoya, Aichi-ken
  - Kitakyushu, Fukuoka
  - Komatsu, Ishikawa-ken
  - Fujisawa, Kanagawa
  - Kawasaki, Kanagawa
  - Sendai, Miyagi
  - Suwa, Nagano
  - Bunkyo-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Chiba
  - Fukuoka
- Mexico (3):
  - Monterrey, Nuevo León
  - Mexico City
  - Querétaro
- Poland (2):
  - Krakow
  - Otwock
- Portugal (2):
  - Coimbra
  - Centro Hospitalar de Lisboa Norte - Hospital Santa Maria, Lisbon
- Russia (2):
  - Novosibirsk
  - Saint Petersburg
- Bratislava, Slovakia
- Seoul, South Korea
- Barcelona, Spain
- Zurich, Switzerland
- Taipei, Taiwan
- Turkey (Türkiye) (3):
  - Ankara
  - Istanbul
  - Izmir
- United Kingdom (2):
  - Cambridge, Cambridgeshire
  - Glasgow, West Dunbartonshire

REFERENCES:
- [Background] Benza RL, Boucly A, Farber HW, Frost AE, Ghofrani HA, Hoeper MM, Lambelet M, Rahner C, Bansilal S, Nikkho S, Meier C, Sitbon O. Change in REVEAL Lite 2 risk score predicts outcomes in patients with pulmonary arterial hypertension in the PATENT study. J Heart Lung Transplant. 2022 Mar;41(3):411-420. doi: 10.1016/j.healun.2021.10.013. Epub 2021 Oct 28. PMID 34848133
- [Background] Benza RL, Farber HW, Frost AE, Ghofrani HA, Corris PA, Lambelet M, Nikkho S, Meier C, Hoeper MM. Application of the REVEAL risk score calculator 2.0 in the CHEST study. Respir Med. 2022 Apr-May;195:106783. doi: 10.1016/j.rmed.2022.106783. Epub 2022 Mar 1. PMID 35256218
- [Derived] Benza RL, Ghofrani HA, Grunig E, Hoeper MM, Jansa P, Jing ZC, Kim NH, Langleben D, Simonneau G, Wang C, Busse D, Meier C, Ghio S. Effect of riociguat on right ventricular function in patients with pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension. J Heart Lung Transplant. 2021 Oct;40(10):1172-1180. doi: 10.1016/j.healun.2021.06.020. Epub 2021 Jul 10. PMID 34353714
- [Derived] Saleh S, Becker C, Frey R, Muck W. Population pharmacokinetics and the pharmacokinetic/pharmacodynamic relationship of riociguat in patients with pulmonary arterial hypertension or chronic thromboembolic pulmonary hypertension. Pulm Circ. 2016 Mar;6(Suppl 1):S86-96. doi: 10.1086/685404. PMID 27162632
- [Derived] Simonneau G, D'Armini AM, Ghofrani HA, Grimminger F, Jansa P, Kim NH, Mayer E, Pulido T, Wang C, Colorado P, Fritsch A, Meier C, Nikkho S, Hoeper MM. Predictors of long-term outcomes in patients treated with riociguat for chronic thromboembolic pulmonary hypertension: data from the CHEST-2 open-label, randomised, long-term extension trial. Lancet Respir Med. 2016 May;4(5):372-80. doi: 10.1016/S2213-2600(16)30022-4. Epub 2016 Apr 8. PMID 27067478
- [Derived] Ghofrani HA, D'Armini AM, Grimminger F, Hoeper MM, Jansa P, Kim NH, Mayer E, Simonneau G, Wilkins MR, Fritsch A, Neuser D, Weimann G, Wang C; CHEST-1 Study Group. Riociguat for the treatment of chronic thromboembolic pulmonary hypertension. N Engl J Med. 2013 Jul 25;369(4):319-29. doi: 10.1056/NEJMoa1209657. PMID 23883377
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 71 centers in 25 countries or regions, between 01-JUL-2009 (first participant first visit) and 19-AUG-2019 (last participant last visit)
Pre-assignment Details: Of the 243 participants who completed CHEST-1 (NCT00855465), 237 entered CHEST-2. 155 participants were from the former riociguat treatment group, and 82 were from the former placebo group.
Groups:
- Riociguat-Former Riociguat 1.0-2.5 mg: Participants were from the former riociguat (BAY 63-2521) treatment group of CHEST-1 on the same dose as they received on the last day of CHEST-1.
- Riociguat-Former Placebo: Participants were from the former placebo group of CHEST-1. The starting dose in CHEST-2 was 1.0 mg riociguat three times one day.
Period: Overall Study
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Started | 155 | 82
Completed | 116 (Completed treatment) | 61 (Completed treatment)
Not Completed | 39 | 21
Not completed — Death | 18 | 12
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Adverse Event | 10 | 5
Not completed — Drug non-compliance | 1 | 0
Not completed — Lack of Efficacy | 4 | 1

BASELINE CHARACTERISTICS:
Population: All 237 participants who completed 16 weeks of treatment in the double-blind CHEST-1 study entered long term extension CHEST-2 study. Baseline of CHEST-2 was Week 0 of CHEST-1. All 237 participants were included in the long-term safety set
Groups:
- Total: Total of all reporting groups
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Total
Number analyzed (Participants) | 155 | 82 | 237
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 91 | 50 | 141
  >=65 years | 64 | 32 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (13.8) | 59.2 (12.4) | 59.1 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 49 | 153
  Male | 51 | 33 | 84
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 105 | 60 | 165
  Black or African American | 7 | 1 | 8
  Asian | 34 | 19 | 53
  Multiple races | 1 | 0 | 1
  Hispanic or Latino | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)
Description: Analyses of drug-related TEAEs were based on the assessment of causal relationship to study medication.
Time Frame: From administration of first dose of study medication up to 2 days after end of treatment with study medication, up to 10 years
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 155 | 82
Participants
  Any TEAE | 153 | 82
  Any drug-related TEAE | 77 | 44
  Any serious TEAE | 96 | 56
  Any drug-related serious TEAE | 14 | 7
  Any TEAT leading to death | 22 | 13

2. Primary Outcome: Number of Participants With Death
Description: Analyses of deaths were based on the assessment of causal relationship to study medication. The safety follow-up visit was to be performed 30 days after the last dose of riociguat.
Time Frame: From baseline to end of safety follow-up visit, up to 10 years (1 month more than End of study visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 155 | 82
Participants | 22 | 13

3. Secondary Outcome: Percentage of Participants With Treatment-emergent High Laboratory Abnormalities in Hematology and Coagulation
Description: Frequency of participants only with a treatment-emergent shift in hematology and coagulation parameters from normal or low at baseline to a high value at a timepoint after the start of treatment. A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to Termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit, and for each parameter.
Measure: Number; unit: Percentage
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 139 | 74
Percentage
  Activated partial thromboplastin time (sec): number analyzed (Participants) | 35 | 21
  Activated partial thromboplastin time (sec) | 97.1 | 90.5
  Basophils (Giga/L): number analyzed (Participants) | 138 | 74
  Basophils (Giga/L) | 1.4 | 0.0
  Basophils / Leukocytes (%): number analyzed (Participants) | 136 | 73
  Basophils / Leukocytes (%) | 18.4 | 16.4
  Eosinophils (Giga/L): number analyzed (Participants) | 137 | 74
  Eosinophils (Giga/L) | 0.7 | 5.4
  Eosinophils / Leukocytes (%): number analyzed (Participants) | 134 | 72
  Eosinophils / Leukocytes (%) | 3.7 | 9.7
  Erythrocytes (T/L): number analyzed (Participants) | 122 | 66
  Erythrocytes (T/L) | 18.0 | 24.2
  Hematocrit (%): number analyzed (Participants) | 85 | 50
  Hematocrit (%) | 41.2 | 38.0
  Hemoglobin (g/dL): number analyzed (Participants) | 128 | 74
  Hemoglobin (g/dL) | 12.5 | 10.8
  Leukocytes (Giga/L): number analyzed (Participants) | 137 | 73
  Leukocytes (Giga/L) | 8.0 | 16.4
  Lymphocytes (Giga/L): number analyzed (Participants) | 139 | 73
  Lymphocytes (Giga/L) | 0.0 | 1.4
  Lymphocytes / Leukocytes (%): number analyzed (Participants) | 136 | 68
  Lymphocytes / Leukocytes (%) | 8.8 | 7.4
  Monocytes (Giga/L): number analyzed (Participants) | 135 | 70
  Monocytes (Giga/L) | 3.7 | 8.6
  Monocytes / Leukocytes (%): number analyzed (Participants) | 135 | 67
  Monocytes / Leukocytes (%) | 15.6 | 16.4
  Neutrophils (Giga/L): number analyzed (Participants) | 133 | 73
  Neutrophils (Giga/L) | 11.3 | 23.3
  Neutrophils / Leukocytes (%): number analyzed (Participants) | 126 | 70
  Neutrophils / Leukocytes (%) | 31.7 | 32.9
  Platelets (Giga/L): number analyzed (Participants) | 122 | 68
  Platelets (Giga/L) | 17.2 | 20.6
  Prothrombin international normalized ratio: number analyzed (Participants) | 26 | 4
  Prothrombin international normalized ratio | 92.3 | 75

4. Secondary Outcome: Percentage of Participants With Treatment-emergent Low Laboratory Abnormalities in Hematology and Coagulation
Description: Frequency of participants only with a treatment-emergent shift in hematology and coagulation parameters from normal or high at baseline to a low value at a timepoint after the start of treatment. A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to Termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit, and for each parameter.
Measure: Number; unit: Percentage
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 139 | 75
Percentage
  Activated partial thromboplastin time (sec): number analyzed (Participants) | 139 | 74
  Activated partial thromboplastin time (sec) | 2.9 | 2.7
  Erythrocytes (T/L): number analyzed (Participants) | 123 | 64
  Erythrocytes (T/L) | 21.1 | 29.7
  Hematocrit (%): number analyzed (Participants) | 129 | 74
  Hematocrit (%) | 9.3 | 17.6
  Hemoglobin (g/dL): number analyzed (Participants) | 120 | 69
  Hemoglobin (g/dL) | 30.0 | 36.2
  Leukocytes (Giga/L): number analyzed (Participants) | 130 | 71
  Leukocytes (Giga/L) | 25.4 | 25.4
  Lymphocytes (Giga/L): number analyzed (Participants) | 130 | 67
  Lymphocytes (Giga/L) | 30.0 | 22.4
  Lymphocytes / Leukocytes (%): number analyzed (Participants) | 112 | 63
  Lymphocytes / Leukocytes (%) | 39.3 | 42.9
  Monocytes (Giga/L): number analyzed (Participants) | 139 | 74
  Monocytes (Giga/L) | 0.7 | 0.0
  Monocytes / Leukocytes (%): number analyzed (Participants) | 139 | 74
  Monocytes / Leukocytes (%) | 3.6 | 2.7
  Neutrophils (Giga/L): number analyzed (Participants) | 139 | 72
  Neutrophils (Giga/L) | 10.8 | 5.6
  Neutrophils / Leukocytes (%): number analyzed (Participants) | 137 | 69
  Neutrophils / Leukocytes (%) | 5.8 | 10.1
  Platelets (Giga/L): number analyzed (Participants) | 131 | 72
  Platelets (Giga/L) | 19.8 | 19.4
  Prothrombin INR: number analyzed (Participants) | 138 | 75
  Prothrombin INR | 0.0 | 0.0

5. Secondary Outcome: Change From Baseline of Hemoglobin in Hematology and Coagulation
Description: Hemoglobin is standard Hematology and coagulation parameter. A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to Termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: gram/deciliter (g/dL)
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 140 | 76
gram/deciliter (g/dL)
  Baseline (Week 0) | 14.49 (1.82) | 14.36 (1.70)
  Change from baseline to Termination visit: number analyzed (Participants) | 5 | 3
  Change from baseline to Termination visit | 1.04 (1.58) | -1.37 (1.71)

6. Secondary Outcome: Percentage of Participants With Treatment-emergent High Laboratory Abnormalities in Clinical Chemistry
Description: Frequency of participants per treatment group only with a treatment-emergent shift in clinical chemistry parameters from normal or low at baseline to a high value at a timepoint after the start of treatment. A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to Termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit, and for each parameter.
Measure: Number; unit: Percentage
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 147 | 77
Percentage
  Alanine aminotransferase (U/L): number analyzed (Participants) | 130 | 73
  Alanine aminotransferase (U/L) | 11.5 | 13.7
  Albumin (g/dL) | 0.0 | 0.0
  Alkaline phosphatase (U/L): number analyzed (Participants) | 127 | 67
  Alkaline phosphatase (U/L) | 22.0 | 19.4
  Aspartate aminotransferase (U/L): number analyzed (Participants) | 134 | 71
  Aspartate aminotransferase (U/L) | 16.4 | 14.1
  Bilirubin (mg/dL): number analyzed (Participants) | 122 | 64
  Bilirubin (mg/dL) | 17.2 | 15.6
  Calcium (mg/dL): number analyzed (Participants) | 38 | 21
  Calcium (mg/dL) | 2.6 | 0.0
  Creatine kinase (U/L): number analyzed (Participants) | 141 | 66
  Creatine kinase (U/L) | 28.4 | 30.3
  Creatinine (mg/dL): number analyzed (Participants) | 83 | 42
  Creatinine (mg/dL) | 32.5 | 31.0
  Gamma glutamyltransferase (U/L): number analyzed (Participants) | 94 | 54
  Gamma glutamyltransferase (U/L) | 22.3 | 24.1
  Glutamate dehydrogenase (U/L): number analyzed (Participants) | 93 | 53
  Glutamate dehydrogenase (U/L) | 43.0 | 34.0
  Phosphate (mg/dL): number analyzed (Participants) | 38 | 20
  Phosphate (mg/dL) | 7.9 | 5.0
  Potassium (mmol/L): number analyzed (Participants) | 141 | 75
  Potassium (mmol/L) | 4.3 | 6.7
  Protein (g/dL): number analyzed (Participants) | 146 | 77
  Protein (g/dL) | 2.7 | 0.0
  Pseudocholinesterase (U/mL): number analyzed (Participants) | 146 | 77
  Pseudocholinesterase (U/mL) | 2.1 | 0.0
  Sodium (mmol/L) | 1.4 | 3.9
  Triacylglycerol lipase (U/L): number analyzed (Participants) | 133 | 69
  Triacylglycerol lipase (U/L) | 18.8 | 18.8
  Urate (mg/dL): number analyzed (Participants) | 110 | 56
  Urate (mg/dL) | 13.6 | 35.7
  Urea (mg/dL): number analyzed (Participants) | 118 | 60
  Urea (mg/dL) | 22.9 | 36.7
  eGFR MDRD method(mL/min/1.73 m2) | 0.0 | 0.0
  Creatinine clearance (mL/min): number analyzed (Participants) | 139 | 70
  Creatinine clearance (mL/min) | 11.5 | 8.6

7. Secondary Outcome: Percentage of Participants With Treatment-emergent Low Laboratory Abnormalities in Clinical Chemistry
Description: Frequency of participants per treatment group only with a treatment-emergent shift in clinical chemistry parameters from normal or high at baseline to a low value at a timepoint after the start of treatment. A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to Termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit, and for each parameter.
Measure: Number; unit: Percentage
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 147 | 77
Percentage
  Albumin (g/dL) | 2.0 | 0.0
  Alkaline phosphatase (U/L): number analyzed (Participants) | 145 | 77
  Alkaline phosphatase (U/L) | 2.1 | 0.0
  Bilirubin (mg/dL): number analyzed (Participants) | 146 | 77
  Bilirubin (mg/dL) | 0.0 | 0.0
  Calcium (mg/dL): number analyzed (Participants) | 35 | 16
  Calcium (mg/dL) | 14.3 | 6.3
  Creatine kinase (U/L): number analyzed (Participants) | 140 | 73
  Creatine kinase (U/L) | 6.4 | 6.8
  Creatinine (mg/dL): number analyzed (Participants) | 146 | 77
  Creatinine (mg/dL) | 4.1 | 3.9
  Gamma glutamyltransferase (U/L) | 0.0 | 0.0
  Phosphate (mg/dL): number analyzed (Participants) | 38 | 21
  Phosphate (mg/dL) | 10.5 | 9.5
  Potassium (mmol/L): number analyzed (Participants) | 141 | 74
  Potassium (mmol/L) | 18.4 | 18.9
  Protein (g/dL): number analyzed (Participants) | 143 | 71
  Protein (g/dL) | 6.3 | 2.8
  Pseudocholinesterase (U/mL): number analyzed (Participants) | 140 | 75
  Pseudocholinesterase (U/mL) | 10.0 | 14.7
  Sodium (mmol/L): number analyzed (Participants) | 141 | 76
  Sodium (mmol/L) | 4.3 | 6.6
  Triacylglycerol lipase (U/L) | 0.0 | 0.0
  Urate (mg/dL): number analyzed (Participants) | 147 | 76
  Urate (mg/dL) | 2.7 | 2.6
  Urea (mg/dL) | 0.0 | 1.3
  eGFR MDRDmethod (mL/min/1.73 m2): number analyzed (Participants) | 105 | 49
  eGFR MDRDmethod (mL/min/1.73 m2) | 26.7 | 22.4
  Creatinine clearance (mL/min): number analyzed (Participants) | 48 | 32
  Creatinine clearance (mL/min) | 29.2 | 40.6

8. Secondary Outcome: Change From Baseline of Urate in Clinical Chemistry
Description: Urate is standard clinical chemistry parameter. A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to Termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 147 | 77
milligram/deciliter (mg/dL)
  Baseline (Week 0) | 6.767 (1.859) | 6.999 (2.193)
  Change from baseline to Termination visit: number analyzed (Participants) | 5 | 3
  Change from baseline to Termination visit | 0.310 (2.916) | -1.290 (1.120)

9. Other Pre Specified Outcome: Change of Systolic Blood Pressure (SBP)
Description: SBP was measured after the participant had been at rest for 10 minutes in a supine position. Low SBP was defined as SBP <95 mmHg, normal SBP as SBP 95-140mmHg, and high SBP as SBP >140 mmHg. A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to Termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: millimetre(s) of mercury (mmHg)
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 155 | 82
millimetre(s) of mercury (mmHg)
  Baseline (Week 0) | 118.81 (14.96) | 124.26 (16.14)
  Change from baseline to Termination visit: number analyzed (Participants) | 126 | 65
  Change from baseline to Termination visit | -3.96 (17.34) | -5.02 (14.79)

10. Other Pre Specified Outcome: Change of Diastolic Blood Pressure (DBP)
Description: DBP was measured after the participants had been at rest for 10 minutes in a supine position. A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to Termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 155 | 82
mmHg
  Baseline (Week 0) | 75.34 (9.75) | 78.55 (9.46)
  Change from baseline to Termination visit: number analyzed (Participants) | 126 | 65
  Change from baseline to Termination visit | -6.16 (13.77) | -7.26 (11.09)

11. Other Pre Specified Outcome: Change of Heart Rate
Description: Heart rate was measured after the participant had been at rest for 10 minutes in a supine position. A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to Termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: beats/minute (BPM)
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 155 | 82
beats/minute (BPM)
  Baseline (Week 0) | 77.66 (12.12) | 76.11 (12.10)
  Change from baseline to Termination visit: number analyzed (Participants) | 126 | 65
  Change from baseline to Termination visit | -0.89 (13.85) | 3.77 (14.69)

12. Other Pre Specified Outcome: Change of Weight
Description: Weight was evaluated for safety. A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to Termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 155 | 82
kilogram (kg)
  Baseline (Week 0) | 74.01 (18.76) | 77.29 (16.42)
  From baseline to Termination visit: number analyzed (Participants) | 123 | 64
  From baseline to Termination visit | -0.87 (5.86) | -2.97 (7.27)

13. Other Pre Specified Outcome: Change of Oxygen Saturation (SaO2)
Description: SaO2 is one parameters of blood gas. The sample was obtained with the participant resting in a sitting or supine position for at least 10 minutes. A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to Termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 154 | 81
Percentage
  Baseline (Week 0) | 93.9 (2.7) | 93.6 (2.4)
  From baseline to Termination visit: number analyzed (Participants) | 3 | 3
  From baseline to Termination visit | 0.0 (2.6) | -2.3 (5.5)

14. Other Pre Specified Outcome: Change of Arterial Partial Oxygen Pressure (PaO2)
Description: PaO2 is one parameter of blood gas. The sample was obtained with the participant resting in a sitting or supine position for at least 10 minutes. A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to Termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 154 | 81
mmHg
  Baseline (Week 0) | 69.66 (11.90) | 69.19 (10.96)
  From baseline to Termination visit: number analyzed (Participants) | 3 | 4
  From baseline to Termination visit | -1.67 (8.02) | 2.00 (24.73)

15. Other Pre Specified Outcome: Change of Arterial Partial Pressure of Carbon Dioxide (PaCO2)
Description: PaCO2 is one parameter of blood gas. The sample was obtained with the participant resting in a sitting or supine position for at least 10 minutes. A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to Termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 154 | 81
mmHg
  Baseline (Week 0) | 33.20 (4.61) | 33.52 (4.60)
  From baseline to Termination visit: number analyzed (Participants) | 3 | 4
  From baseline to Termination visit | -0.33 (1.53) | -2.25 (4.5)

16. Other Pre Specified Outcome: Change of RR Duration From Electrocardiogram (ECG)
Description: Heart rate from ECG is derived from the RR duration, unless arrhythmias such as atrial fibrillation or ventricular extra beats require additional calculations. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position. Analyses up to Month 48. After this timepoint, data was available for considerably fewer participants in the analysis set.
Time Frame: From baseline to Month 48
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 149 | 75
millisecond (msec)
  Baseline (Week 0) | 812.90 (144.31) | 828.47 (147.54)
  Change rom baseline to Month 48: number analyzed (Participants) | 2 | 0
  Change rom baseline to Month 48 | 152.00 (236.17) |

17. Other Pre Specified Outcome: Change of PR Duration From ECG
Description: PR duration was evaluated as part of ECG. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position. Analyses up to Month 48. After this timepoint, data was available for considerably fewer participants in the analysis set.
Time Frame: From baseline to Month 48
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 147 | 72
msec
  Baseline (Week 0) | 173.22 (26.49) | 174.92 (24.35)
  Change from baseline to Month 48: number analyzed (Participants) | 2 | 0
  Change from baseline to Month 48 | -10.00 (11.31) |

18. Other Pre Specified Outcome: Change of QRS Duration From ECG
Description: QRS duration was evaluated as part of ECG. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position. Analyses up to Month 48. After this timepoint, data was available for considerably fewer participants in the analysis set.
Time Frame: From baseline to Month 48
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 148 | 74
msec
  Baseline (Week 0) | 104.30 (17.85) | 104.11 (18.24)
  Change from baseline to Month 48: number analyzed (Participants) | 2 | 0
  Change from baseline to Month 48 | 3.00 (4.24) |

19. Other Pre Specified Outcome: Change of QT Duration in ECG
Description: QT duration was evaluated as part of ECG. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position. Analyses up to Month 48. After this timepoint, data was available for considerably fewer participants in the analysis set.
Time Frame: From baseline to Month 48
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 114 | 53
msec
  Baseline (Week 0) | 405.82 (31.29) | 408.45 (30.98)
  Change from baseline to Month 48: number analyzed (Participants) | 2 | 0
  Change from baseline to Month 48 | 42.00 (39.60) |

20. Other Pre Specified Outcome: Change in Six-minute Walking Distance (6MWD) Test
Description: 6MWD is exercise testing and is one of efficacy evaluation
Time Frame: From baseline to End of study visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Median (Full Range); unit: meters
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 155 | 82
meters
  Baseline (Week 0) | 361.0 [150 to 557] | 372.0 [170 to 474]
  Change from baseline to End of study visit | 31.0 [-447 to 230] | 12.5 [-448 to 215]

21. Other Pre Specified Outcome: Change in Pulmonary Vascular Resistance (PVR)
Description: Pulmonary vascular resistance (PVR) was measured only if right-heart catheterization was performed as part of a regular diagnostic work-up. Analyses up to Month 48 due to limited data.
Time Frame: From baseline to Month 45 and Month 48
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: dyn*s*cm^-5
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 146 | 80
dyn*s*cm^-5
  Baseline (Week 0) | 796.64 (435.24) | 761.83 (388.87)
  Change from baseline to Month 45: number analyzed (Participants) | 0 | 1
  Change from baseline to Month 45 |  | -1243.48 (NA) — The value was not calculated due to very low number of participants
  Change from baseline to Month 48: number analyzed (Participants) | 2 | 0
  Change from baseline to Month 48 | -148.29 (74.39) |

22. Other Pre Specified Outcome: Change in N-terminal Prohormone of Brain Natriuretic Peptide (NT-proBNP)
Description: NT-proBNP levels in the blood are used for diagnosis of acute congestive heart failure (CHF) and may be useful to establish prognosis in heart failure
Time Frame: From baseline to End of study visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: picograms/millilitre (pg/mL)
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 135 | 69
picograms/millilitre (pg/mL)
  Baseline (Week 0) | 1553.19 (2435.94) | 1404.23 (1745.48)
  Change from baseline to End of study visit | -125.99 (2503.78) | -187.96 (1438.96)

23. Other Pre Specified Outcome: Change in World Health Organization (WHO) Functional Class
Description: WHO classification: I: Participants with PH. Ordinary physical activity does not cause undue dyspnea or fatigue, chest pain, or near syncope. II: Participants with PH are comfortable at rest. Ordinary physical activity causes undue dyspnea or fatigue, chest pain, or near syncope. III: Participants with PH are comfortable at rest. Less than ordinary activity causes undue dyspnea or fatigue, chest pain, or near syncope. IV: Participants with PH with inability to carry out any physical activity. They manifest signs of right-heart failure. Dyspnea and/or fatigue may even be present at rest. For class change from baseline, minus indicates a participant's functional class decreased compared with baseline (e.g. "-1" indicates a participant changed from class IV to class III, or from class II to class I), plus indicates a participant's functional class increased compared with baseline (e.g. "+1" indicates a participant changed from class I to class II, or from class III to class IV).
Time Frame: From baseline to End of study visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 155 | 82
Participants
  Baseline (Week 0)-class I | 3 | 0
  Baseline (Week 0)-class II | 48 | 25
  Baseline (Week 0)-class III | 100 | 54
  Baseline (Week 0)-class IV | 4 | 2
  Baseline (Week 0)-Missing | 0 | 1
  Change from baseline to End of study visit- -2: number analyzed (Participants) | 155 | 81
  Change from baseline to End of study visit- -2 | 7 | 4
  Change from baseline to End of study visit- -1: number analyzed (Participants) | 155 | 81
  Change from baseline to End of study visit- -1 | 44 | 24
  Change from baseline to End of study visit- -0: number analyzed (Participants) | 155 | 81
  Change from baseline to End of study visit- -0 | 72 | 38
  Change from baseline to End of study visit- +1: number analyzed (Participants) | 155 | 81
  Change from baseline to End of study visit- +1 | 11 | 2
  Change from baseline to End of study visit- +2: number analyzed (Participants) | 155 | 81
  Change from baseline to End of study visit- +2 | 13 | 7
  Change from baseline to End of study visit- +3: number analyzed (Participants) | 155 | 81
  Change from baseline to End of study visit- +3 | 7 | 6
  Change from baseline to End of study visit- +4: number analyzed (Participants) | 155 | 81
  Change from baseline to End of study visit- +4 | 1 | 0

24. Other Pre Specified Outcome: Number of Participants With Clinical Worsening
Description: Time to clinical worsening was a parameter that combined death and events reflective of persistent clinical worsening of the participant's underlying diagnosis of pulmonary hypertension (PH).
Time Frame: From baseline to End of study visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 155 | 82
Participants
  Any clinical worsening | 45 | 23
  Pulmonary endarterectomy | 4 | 3
  Hospitalization due to PH | 7 | 3
  Start of new PH treatment | 21 | 9
  Decrease in 6MWD due to PH | 4 | 2
  Persistent worsening of functional class due to PH | 7 | 2
  Death | 22 | 13

25. Other Pre Specified Outcome: Incidence of Clinical Worsening Events Per 100 Person Years
Description: as for outcome 24
Time Frame: From baseline to End of study visit, up to 10 years
Measure: Number; unit: Percentage per 100 person-years
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 155 | 82
Percentage per 100 person-years
  Any clinical worsening event | 12.84 | 11.77
  Pulmonary endarterectomy | 0.73 | 1.04
  Hospitalization due to PH | 1.65 | 1.04
  Start of new PH treatment | 4.40 | 3.81
  Decrease in 6MWD due to PH | 0.73 | 0.69
  Persistent worsening of functional class due to PH | 1.28 | 0.69
  Death | 4.04 | 4.50

26. Other Pre Specified Outcome: Change From Baseline in Borg CR 10 Scale
Description: The Borg CR10 Scale was measured in conjunction with the 6MWD test. The test was explained to the participant before starting the 6MWD test. Participants were asked to rank their exertion at the end of the 6MWD test. Low values indicate low levels of exertion; high values indicate more intense exertion reported by the participant. The score ranges from 0 ("Nothing at all") to 10 ("Extremely strong - Maximal").
Time Frame: From baseline to Week 12
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 155 | 82
Scores on a scale
  Baseline (Week 0) | 4.36 (2.30) | 4.45 (2.26)
  Change from baseline to Week 12 | -0.93 (2.47) | -0.3 (2.08)

27. Other Pre Specified Outcome: Change in Score of EQ-5D Questionnaire
Description: The EQ-5D is a standardized instrument for use as a measure of health outcome. The EQ-5D is a self report questionnaire. The utility score is calculated based on five questions concerning problems with mobility, self-care, usual activities, pain/discomfort and anxiety/depression. An increase in the utility score represents an improvement in quality of life. The score ranges from -0.594 (worst answer in all five questions) to 1 (best answer in all five questions).
Time Frame: From baseline to End of study visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 154 | 81
Scores on a scale
  Baseline (Week 0) | 0.6406 (0.2509) | 0.6569 (0.2518)
  Change from baseline to EOS Visit | -0.1008 (0.4965) | -0.1230 (0.5213)

28. Other Pre Specified Outcome: Change in Score of Living With Pulmonary Hypertension (LPH) Questionnaire
Description: The LPH questionnaire is designed to measure the effects of PH and PH-specific treatments on an individual's quality of life. The LPH is a self-report questionnaire and was completed by the participant. The LPH total score can range from 0 (best) to 105 (worst).
Time Frame: From baseline to End of study visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo
Number analyzed (Participants) | 152 | 80
Scores on a scale
  Baseline (Week 0) | 42.19 (22.05) | 46.01 (22.93)
  Change from baseline to EOS Visit | -2.64 (29.26) | -0.56 (30.83)

ADVERSE EVENTS:
Time Frame: From administration of first dose of study medication up to 2 days after end of treatment with study medication, up to 10 years.
Groups:
- Former Riociguat 1.0-2.5 mg: Subjects from the riociguat 1.0-2.5 mg group of CHEST-1 entered the extension study(CHEST-2) with the same dose as they received on the last day of CHEST-1 (Visit7).
- Former Placebo: Subjects from the placebo group of CHEST-1 entered the extension study (CHEST-2),the starting dose in CHEST-2 was 1.0 mg riociguat tid.
Arm/Group | Former Riociguat 1.0-2.5 mg | Former Placebo
All-Cause Mortality (participants affected / at risk) | 22/155 | 13/82
Serious Adverse Events (participants affected / at risk) | 96/155 | 56/82
Other Adverse Events (participants affected / at risk) | 148/155 | 79/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Former Riociguat 1.0-2.5 mg (N=155) | Former Placebo (N=82)
Anaemia (Blood and lymphatic system disorders) | 4 (6) | 2 (2)
Bicytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 5 (6)
Atrial flutter (Cardiac disorders) | 5 (7) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 5 (5) | 2 (2)
Cardiac failure (Cardiac disorders) | 8 (9) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Cor pulmonale chronic (Cardiac disorders) | 1 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 13 (24) | 8 (13)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute right ventricular failure (Cardiac disorders) | 3 (6) | 0 (0)
Myxoedema (Endocrine disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (5) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (3) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (7) | 3 (4)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (2) | 2 (3)
Death (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 2 (2)
Pelvic mass (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (2) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (3) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (3)
Infection (Infections and infestations) | 2 (3) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (2)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 17 (20) | 7 (8)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (5)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (2)
Subdiaphragmatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Bone abscess (Infections and infestations) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Angiogram pulmonary (Investigations) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Catheterisation cardiac (Investigations) | 8 (9) | 3 (3)
Colonoscopy (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Investigation (Investigations) | 2 (2) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Steroid diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 14 (16) | 11 (17)
Vertebrobasilar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Psychiatric decompensation (Psychiatric disorders) | 1 (1) | 0 (0)
Vascular cognitive impairment (Psychiatric disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 5 (6)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 16 (29) | 13 (15)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Angioplasty (Surgical and medical procedures) | 0 (0) | 2 (4)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Colostomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Peritoneal dialysis (Surgical and medical procedures) | 1 (1) | 0 (0)
Removal of internal fixation (Surgical and medical procedures) | 0 (0) | 1 (1)
Splenectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Vitrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Vena cava filter insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Cervical conisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 0 (0) | 1 (1)
Pulmonary artery therapeutic procedure (Surgical and medical procedures) | 0 (0) | 1 (5)
Cataract operation (Surgical and medical procedures) | 1 (2) | 0 (0)
Pulmonary endarterectomy (Surgical and medical procedures) | 2 (2) | 3 (3)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Temporal arteritis (Vascular disorders) | 1 (2) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (4)
Device dislocation (Product Issues) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Former Riociguat 1.0-2.5 mg (N=155) | Former Placebo (N=82)
Anaemia (Blood and lymphatic system disorders) | 15 (24) | 9 (9)
Atrial fibrillation (Cardiac disorders) | 12 (13) | 6 (11)
Palpitations (Cardiac disorders) | 13 (15) | 9 (11)
Supraventricular extrasystoles (Cardiac disorders) | 2 (3) | 5 (8)
Ventricular extrasystoles (Cardiac disorders) | 4 (4) | 5 (8)
Abdominal pain (Gastrointestinal disorders) | 8 (11) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 13 (16) | 7 (9)
Constipation (Gastrointestinal disorders) | 14 (17) | 9 (11)
Diarrhoea (Gastrointestinal disorders) | 30 (37) | 17 (27)
Dyspepsia (Gastrointestinal disorders) | 17 (22) | 11 (12)
Gastritis (Gastrointestinal disorders) | 4 (5) | 6 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 (10) | 4 (5)
Nausea (Gastrointestinal disorders) | 19 (23) | 16 (27)
Toothache (Gastrointestinal disorders) | 10 (10) | 4 (4)
Vomiting (Gastrointestinal disorders) | 15 (19) | 8 (8)
Chest discomfort (General disorders) | 7 (12) | 7 (9)
Chest pain (General disorders) | 15 (20) | 8 (10)
Fatigue (General disorders) | 10 (10) | 8 (8)
Oedema (General disorders) | 6 (8) | 8 (13)
Oedema peripheral (General disorders) | 38 (58) | 27 (40)
Pyrexia (General disorders) | 9 (11) | 4 (7)
Bronchitis (Infections and infestations) | 24 (39) | 11 (15)
Influenza (Infections and infestations) | 7 (7) | 5 (8)
Nasopharyngitis (Infections and infestations) | 55 (108) | 24 (47)
Pneumonia (Infections and infestations) | 11 (12) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 26 (32) | 13 (25)
Urinary tract infection (Infections and infestations) | 15 (24) | 9 (15)
Respiratory tract infection (Infections and infestations) | 12 (27) | 8 (17)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
Ligament sprain (Injury, poisoning and procedural complications) | 9 (10) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 12 (16) | 7 (8)
Activated partial thromboplastin time prolonged (Investigations) | 10 (15) | 2 (2)
Blood potassium decreased (Investigations) | 1 (1) | 5 (9)
International normalised ratio increased (Investigations) | 13 (19) | 6 (6)
Hyperuricaemia (Metabolism and nutrition disorders) | 5 (5) | 7 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 16 (20) | 9 (14)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 (33) | 10 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (40) | 11 (14)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (12) | 4 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (16) | 8 (11)
Dizziness (Nervous system disorders) | 34 (47) | 20 (28)
Headache (Nervous system disorders) | 14 (19) | 12 (21)
Insomnia (Psychiatric disorders) | 8 (8) | 9 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (34) | 17 (23)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 (29) | 15 (23)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 (20) | 11 (15)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 6 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 9 (10)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 3 (4)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 8 (16) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (10) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6)
Hypotension (Vascular disorders) | 12 (13) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2012-12-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT00910429/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT00910429/SAP_001.pdf